CLINICAL TRIAL: NCT04128514
Title: Spectacle Independence and Overall Satisfaction With Bilateral Implantation of the AcrySof® Panoptix® Toric Intraocular Lens
Brief Title: Spectacle Independence and Overall Satisfaction With AcrySof® Panoptix® Toric Intraocular Lens
Status: Terminated | Type: Observational
Why Stopped: Insufficient enrollment
Sponsor: Eye Center of North Florida (Other)
Collaborators: Science in Vision (Other)
Responsible Party: Sponsor
Other Study IDs: BF-19-001
Record Dates: First submitted 2019-10-10; First posted 2019-10-16 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Cataract
Keywords: Toric IOL; Panoptix; multifocal IOL; trifocal IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Enrolled subjects: Subjects ≥40 years of age presenting for cataract surgery who are interested in reducing their dependence on spectacles at all distances, and who are appropriate candidates for multifocal lens implantation.
  The Acrysof (R) Panoptix (R) Toric intraocular lens will be implanted in both eyes of subjects.
  Interventions: Device: Panoptix Toric

INTERVENTIONS:
Device: Panoptix Toric — Cataract surgery and IOL implantation

SUMMARY:
The study was designed to assess the spectacle independence and satisfaction of patients receiving the AcrySof® Panoptix® Toric intraocular lens (IOL) after uneventful cataract surgery.

DETAILED DESCRIPTION:
This study is a single-arm unmasked clinical evaluation study of spectacle independence after successful bilateral cataract surgery. Subjects will be assessed pre-operatively, operatively and at 1 day, 1 month and 3 months post-operatively. Clinical evaluations will include administration of a spectacle independence and a quality of life questionnaire, as well as measurement of bilateral visual acuity and manifest refraction.

ELIGIBILITY:
Inclusion Criteria

Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

* Presenting for uncomplicated bilateral cataract surgery and have an interest in spectacle independence using a multifocal toric IOL option
* Gender: Males and Females.
* Age: 40 or older.
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.
* Have good ocular health, with no pathology that compromises visual acuity (outside of residual refractive error and cataract)
* Have regular corneal astigmatism with a magnitude that can be treated with a toric IOL in the approved range (T3-T6) for the Panoptix lens.
* Have 20/32 (0.2 logMAR) or better potential acuity in both eyes

Exclusion Criteria If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Irregular astigmatism (e.g. keratoconus)
* Corneal pathology (e.g. scar, dystrophy, pterygium, moderate-to-severe dry eye)
* Monocular status (e.g. amblyopia)
* Previous radial keratotomy, corneal refractive surgery or other corneal surgery (e.g. corneal transplant, DSAEK, lamellar keratoplasty)
* Previous anterior or posterior chamber surgery (e.g., vitrectomy, laser iridotomy)
* Diabetic retinopathy
* Macular pathology (e.g. ARMD, ERM)
* History of retinal detachment
* Subjects who have an acute or chronic disease or illness that would confound the results of this investigation (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness), that are known to affect postoperative visual acuity.
* Participation in any investigational drug or device trial within the previous 30 days prior to the start date of this trial (or currently participating).

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects ≥40 years of age presenting for cataract surgery who are interested in reducing their dependence on spectacles at all distances, and who are appropriate candidates for multifocal lens implantation.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Spectacle independence - emmetropia | 3 months
  Percent of patients with ≤ 0.5D of refractive cylinder and ≤ 0.50D of absolute residual spherical equivalent refraction postoperatively who never or rarely wear spectacles for distance, intermediate or near vision 3 months postop (based on the Patient-Reported Spectacle Independence Questionnaire, or PRSIQ1 - "a little of the time" or "none of the time")

SECONDARY OUTCOMES:
Binocular uncorrected distance visual acuity | 3 months
  Binocular distance visual acuity
Binocular uncorrected intermediate visual acuity | 3 months
  Binocular intermediate visual acuity
BInocular uncorrected near visual acuity | 3 months
  Binocular near visual acuity
Binocular best-corrected distance visual acuity | 3 months
  Binocular best-corrected distance visual acuity
Binocular distance-corrected intermediate visual acuity | 3 months
  Binocular distance-corrected intermediate visual acuity
Binocular distance-corrected near visual acuity | 3 months
  Binocular distance-corrected near visual acuity
Spherical equivalent refraction | 3 months
  Spherical equivalent refraction
Residual astigmatism | 3 months
  Residual astigmatism
Uncorrected preferred reading distance | 3 months
  Uncorrected preferred reading distance
Monocular corrected distance visual acuity | 3 months
  Monocular corrected distance visual acuity
Spectacle independence - overall | 3 months
  Percent of all patients who never or rarely wear spectacles for distance, intermediate or near vision 3 months postop (based on the Patient-Reported Spectacle Independence Questionnaire, or PRSIQ1 - "a little of the time" or "none of the time")
Binocular uncorrected visual acuity at preferred reading distance | 3 months
  Binocular uncorrected visual acuity at preferred reading distance
VFQ-14 | 3 months
  Questionnaire responses on VFQ-14 visual function questionnaire
Choose lens again | 3 months
  Percent of patients who would choose this lens modality again.

CONTACTS AND LOCATIONS:
Overall Officials: Bret Fisher, MD, Principal Investigator — Eye Center of North Florida
Locations (1):
- Eye Center of North Florida, Panama City, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
No current plans to share data, but if shared, any shared outcomes data will be de-identified before release.

REFERENCES:
- [Background] Morlock R, Wirth RJ, Tally SR, Garufis C, Heichel CWD. Patient-Reported Spectacle Independence Questionnaire (PRSIQ): Development and Validation. Am J Ophthalmol. 2017 Jun;178:101-114. doi: 10.1016/j.ajo.2017.03.018. Epub 2017 Mar 22. PMID 28341605
- [Background] Akman A, Asena L, Ozturk C, Gur Gungor S. Evaluation of quality of life after implantation of a new trifocal intraocular lens. J Cataract Refract Surg. 2019 Feb;45(2):130-134. doi: 10.1016/j.jcrs.2018.12.003. Epub 2019 Jan 3. PMID 30612749